CLINICAL TRIAL: NCT01023802
Title: The Use of Molecular Breast Imaging in the Evaluation of Tumor Response to Neoadjuvant Therapy in Women With Breast Cancer - A Pilot Study
Brief Title: The Use of Molecular Breast Imaging in the Evaluation of Tumor Response to Neoadjuvant Therapy in Women With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, M.D., Mayo Clinic
Other Study IDs: 09-005183
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Neoadjuvant Therapy; Chemotherapy; Hormone Replacement Therapy; Breast Cancer
Keywords: neoadjuvant therapy; chemotherapy; hormone therapy; breast cancer; MBI; Molecular Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neoadjuvant therapy for breast cancer: Women who present to the Internal Medicine Breast Cancer Clinic with breast cancer and who after discussion with the consulting surgeon and oncologist have agreed to undergo neoadjuvant chemotherapy or neoadjuvant hormone therapy.

SUMMARY:
In patients with breast cancer who undergo neoadjuvant chemotherapy or neoadjuvant hormone therapy molecular breast imaging (MBI) is an accurate test for assessing response rate to neoadjuvant therapy.

DETAILED DESCRIPTION:
The investigators propose to evaluate Molecular Breast Imaging in patients undergoing neoadjuvant therapy for breast cancer with the aims to document that 1) the change in uptake of 99mTc-sestamibi prior to initiation of neoadjuvant therapy, after 3-5 weeks of neoadjuvant therapy and at completion of neoadjuvant therapy prior to breast cancer surgery will be a reflection of the tumor response to neoadjuvant therapy.

2) Tumor response at 3-5 weeks of neoadjuvant therapy is predictive of tumor response at completions of neoadjuvant therapy.

3) Post-neoadjuvant tumor size as determined by MBI corresponds to size found at surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer scheduled to undergo neoadjuvant chemotherapy therapy or neoadjuvant hormone therapy and who have undergone any breast imaging procedure, and in whom a repeat imaging procedure is planned prior to definite surgery. MRI of the breast for accurate tumor size evaluation is recommended but not necessarily required for study inclusion.
* Are able to return for a 3-5 week follow-up MBI study and for the final MBI study at completion of the neoadjuvant therapy.
* Patient age > 18

Exclusion Criteria:

* Unable to understand or sign a consent form
* Pregnant or lactating
* Physically unable to sit upright and still for 40 minutes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients who present to the Internal Medicine Breast Cancer Clinic with breast cancer and who after discussion with the consulting surgeon and oncologist have agreed to undergo neoadjuvant chemotherapy or neoadjuvant hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic You Tude Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/